CLINICAL TRIAL: NCT06406127
Title: Effect of Alpha Lipoic Acid on Chemotherapy Induced Neurological Changes in Breast Cancer Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Dar EL Salam Cancer Hospital (Unknown)
Responsible Party: Principal Investigator, Shaimaa Mohamed SafaaElDin, Pharmacist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RHDIRB2020110301 REC #247
Record Dates: First submitted 2024-04-19; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Alpha Lipoic Acid; Paclitaxel; Neurologic Disorder; Chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Nervous System Diseases | interventions — Thioctic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy + Alpha Lipoic Acid (Experimental): will receive chemotherapy (paclitaxel for 12 weeks) + Alpha Lipoic Acid for 14 weeks (one week before the start of paclitaxel and continue for one week after the end of paclitaxel).
  Interventions: Drug: Alpha Lipoic Acid 600 MG Oral Capsule
- Chemotherapy only (No Intervention): will receive chemotherapy only (paclitaxel for 12 weeks).

INTERVENTIONS:
Drug: Alpha Lipoic Acid 600 MG Oral Capsule — Single 600 mg daily dose
  Other Names: No drug
  Arms: Chemotherapy + Alpha Lipoic Acid

SUMMARY:
92 female cancer patients, aged from 18 to 75 years old (with a first diagnosis of breast cancer) who will receive Paclitaxel-based chemotherapy (12 weeks) as first line therapy, will be enrolled in the study and will be randomly assigned to either:

* Group I: will receive the chemotherapy protocol or
* Group II: will receive the chemotherapy protocol plus 600 mg daily dose of Alpha Lipoic Acid for 14 weeks (one week before the start of paclitaxel and continue till one week after the end of paclitaxel).

  * Blood samples will be withdrawn 2 times (week 1 and week 12) to measure the following: (Stored in -80 C till the end of the study)
* Tumor Necrotizing Factor- alpha (TNF-α) by ELISA.
* Brain-Derived Neurotrophic Factor (BDNF) by ELISA.

  * All patients will be subjected to 6 tests/questionnaires (week 1 - week 12 - week 24) to predict the functionality of the brain:
* Functional Assessment of Cancer Therapy-Cognitive (FACT-Cog) version 3
* Mini-Cog Test
* Mini Mental State Examination (MMSE)
* Controlled Oral Word Association Test (COWAT)
* Hopkins Verbal Learning Test (HVLT)
* Trail Making Test (TMT)

DETAILED DESCRIPTION:
92 Female Cancer patients will be randomized to 2 groups, the first group will receive the alpha lipoic acid beside their chemotherapy regimen and the other group will only receive the chemotherapy regimen. Both groups will be watched for any changes in their neurological behaviors by asking and receiving answers on the questionnaires that were mentioned before. This will be done in 3 different time margins:

* Before starting the chemotherapeutic regimen
* after ending the chemotherapeutic regimen
* after 6 months of receiving the chemotherapeutic regimen this will show even the late symptoms and effects of the chemotherapy. Also serum biomarkers will be measured (TNF alpha and BDNF) 2 times; one before starting the chemotherapeutic regimen and the other after ending the treatment.

Throughout the treatment process, both groups will be monitored for any side effects concerning the alpha lipoic acid or the chemotherapeutic regimen.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer patients aged 18 to 75 years old.
* Patients with a first diagnosis of cancer and indication for first-line therapy with Paclitaxel-based chemotherapy.
* Patients are those who are diagnosed with Stage 1 to 3 non-metastatic breast cancer.
* Patients are intended to receive 12 weeks of paclitaxel (75 - 80 mg/m2) according to the TC protocol.
* No previous neurological conditions (including dementia, Alzheimer's disease, Parkinson's disease) and taking no neurological-related drugs.
* Normal hepatic and renal function (bilirubin ≤1.5 mg/dL, creatinine ≤2.0 mg/dL).
* Eastern Cooperative Oncology Group (ECOG) performance status from 0 - 2.
* Patient Health Questionnaire (PHQ) score from 0 - 9.

Exclusion Criteria:

* Hypersensitivity / Allergy to Alpha Lipoic Acid.
* Any condition that contraindicates chemotherapy (i.e., pregnancy, lactation).
* New-onset neurological symptoms or presence of any neurological disorder.
* Patients with known history or current treatment with neurological agents.
* Alcohol abuse.
* Current participation in any other clinical investigation.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Tumor Necrotizing Factor Alpha Serum Levels | At baseline of treatment and After 12 weeks of the paclitaxel-based therapy (at the end of therapy)
  All patients will be evaluated during the trial for 2 times via monitoring the Tumor Necrotizing Factor- alpha (TNF-α).

SECONDARY OUTCOMES:
Response assessment by questionnaire - FACT-COG Test | For 3 times during the study: - At baseline - After 12 weeks of the paclitaxel-based therapy. - After 6 months from the start of the paclitaxel-based therapy.
  Evaluation of response will be done guided by the questionnaire to detect the neuropsychiatric panel.
  FACT Cognitive function version 3 consists of questions regarding:
  * Perceived cognitive impairments.
  * Comments from others.
  * Perceived cognitive abilities.
  * Impact on quality of life. For every answered question, the patient receives points on a scale of scores. Those scales will be compared in every time the questionnaire is conducted to assess the functionality of the brain.
  The scale of numbers of the answers is:
  * Never = 0
  * About once a week = 1
  * Two to three times a week = 2
  * Nearly every day = 3
  * Several times a day = 4 It is better when the patient has low score.
Response assessment by questionnaire - Mini-Cog Test | For 3 times during the study: - At baseline - After 12 weeks of the paclitaxel-based therapy. - After 6 months from the start of the paclitaxel-based therapy.
  Evaluation of response will be done guided by the questionnaire to detect the neuropsychiatric panel.
  Mini-Cog Test consists of three steps:
  * Three Word Registration: Telling the patient a list of words and ask him to memorize them.
  * Clock Drawing: Asking the patient to draw the clock and record the time taken for drawing. Normal clock = 2 points. Inability or refusal to draw a clock (abnormal) = 0 points.
  * Three-Word Recall: Asking the patient to recall the list of words done in step 1.
  For every word recalled, patient receives a point. Total points will be compared in every time the questionnaire is done to assess the functionality of the brain.
Response assessment by questionnaire - Mini Mental State Examination (MMSE) | For 3 times during the study: - At baseline - After 12 weeks of the paclitaxel-based therapy. - After 6 months from the start of the paclitaxel-based therapy.
  Evaluation of response will be done guided by the questionnaire to detect the neuropsychiatric panel.
  MMSE consists of questions regarding:
  * Orientation to time (2 points, one for each question)
  * Orientation to place (2 points, one for each question)
  * Concentration and attention (2 questions and for each question this scale will be applied: No Errors - 2 points, 1 Error - 1 point, 2 or more Errors - 0 points)
  * Delayed recall (3 points, one for each recalled word) For every answered question, the patient will get points. Those points will be compared in every phase the questionnaire is done for every patient.
Response assessment by questionnaire - Controlled Oral Word Association Test (COWAT) | For 3 times during the study: - At baseline - After 12 weeks of the paclitaxel-based therapy. - After 6 months from the start of the paclitaxel-based therapy.
  Evaluation of response will be done guided by the questionnaire to detect the neuropsychiatric panel.
  The patient is asked to tell words that begin with a certain alphabet in a certain time margin. This will be done for 4 different alphabets and words will be recorded to calculate the score.
  Points of every alphabet will be compared in every time the questionnaire is conducted to assess the functionality of the brain.
  The more words told in the same time margin, the better.
Response assessment by questionnaire - The Verbal Memory Arabic Test (VMAT) | For 3 times during the study: - At baseline - After 12 weeks of the paclitaxel-based therapy. - After 6 months from the start of the paclitaxel-based therapy.
  Evaluation of response will be done guided by the questionnaire to detect the neuropsychiatric panel.
  The VMAT consists of 3 trials of delayed recall. Every trial has a list of words for which the patient will be asked to recall. For every recalled word the patient will have a point and those points will be compared in every time the questionnaire is conducted to assess the functionality of the brain.
  The more words recalled, the better.
Response assessment by questionnaire - Trail Making Test (TMT) | For 3 times during the study: - At baseline - After 12 weeks of the paclitaxel-based therapy. - After 6 months from the start of the paclitaxel-based therapy.
  Evaluation of response will be done guided by the questionnaire to detect the neuropsychiatric panel.
  TMT consists of 2 parts, A and B. Both parts of the Trail Making Test consist of 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers and letters; as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.).
  Results for both TMT A and B are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
Brain Derived Neurotrophic Factor Serum Levels | At baseline and After 12 weeks of the paclitaxel-based therapy (at the end of therapy)
  All patients will be evaluated during the trial for 2 times via monitoring Brain-Derived Neurotrophic Factor (BDNF) serum levels.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | through study completion, an average of 1 year.
  Monitoring alpha lipoic acid related adverse reactions:
  Headache, heartburn, nausea and vomiting are nearly the most common adverse effects concerning alpha lipoic acid.
Monitoring the chemotherapy toxicity and side effects. | through study completion, an average of 1 year.
  National Cancer Institute common Terminology criteria for Adverse Effect grading: NCI-CTCAE version 4.0. for evaluation of chemotherapy toxicities.
Monitoring Drug-Drug interactions. | through study completion, an average of 1 year.
  Including chemotherapeutic agents and any other add-on medication.

CONTACTS AND LOCATIONS:
Overall Officials: Manal H El Hamamsy, Doctorate, Principal Investigator — Ain Shams University - Faculty of Pharmacy
Locations (1):
- Dar El Salam Cancer Hospital (Harmel Hospital), Cairo, El Malek El Saleh, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] NCD Countdown 2030 collaborators. NCD Countdown 2030: worldwide trends in non-communicable disease mortality and progress towards Sustainable Development Goal target 3.4. Lancet. 2018 Sep 22;392(10152):1072-1088. doi: 10.1016/S0140-6736(18)31992-5. Epub 2018 Sep 20. PMID 30264707
- [Result] Rostom Y, Abdelmoneim SE, Shaker M, Mahmoud N. Presentation and management of female breast cancer in Egypt. East Mediterr Health J. 2022 Oct 30;28(10):725-732. doi: 10.26719/emhj.22.076. PMID 36382727
- [Result] Brown T, McElroy T, Simmons P, Walters H, Ntagwabira F, Wang J, Byrum SD, Allen AR. Cognitive impairment resulting from treatment with docetaxel, doxorubicin, and cyclophosphamide. Brain Res. 2021 Jun 1;1760:147397. doi: 10.1016/j.brainres.2021.147397. Epub 2021 Mar 8. PMID 33705788
- [Result] Bellens A, Roelant E, Sabbe B, Peeters M, van Dam PA. A video-game based cognitive training for breast cancer survivors with cognitive impairment: A prospective randomized pilot trial. Breast. 2020 Oct;53:23-32. doi: 10.1016/j.breast.2020.06.003. Epub 2020 Jun 12. PMID 32554133
- [Result] Janelsins MC, Kohli S, Mohile SG, Usuki K, Ahles TA, Morrow GR. An update on cancer- and chemotherapy-related cognitive dysfunction: current status. Semin Oncol. 2011 Jun;38(3):431-8. doi: 10.1053/j.seminoncol.2011.03.014. PMID 21600374
- [Result] Lee JH, Nan A. Combination drug delivery approaches in metastatic breast cancer. J Drug Deliv. 2012;2012:915375. doi: 10.1155/2012/915375. Epub 2012 Apr 26. PMID 22619725
- [Result] Emadi A, Jones RJ, Brodsky RA. Cyclophosphamide and cancer: golden anniversary. Nat Rev Clin Oncol. 2009 Nov;6(11):638-47. doi: 10.1038/nrclinonc.2009.146. Epub 2009 Sep 29. PMID 19786984
- [Result] Inagaki M, Yoshikawa E, Matsuoka Y, Sugawara Y, Nakano T, Akechi T, Wada N, Imoto S, Murakami K, Uchitomi Y. Smaller regional volumes of brain gray and white matter demonstrated in breast cancer survivors exposed to adjuvant chemotherapy. Cancer. 2007 Jan 1;109(1):146-56. doi: 10.1002/cncr.22368. PMID 17131349
- [Result] Schultz C, Engelhardt M. Anatomy of the hippocampal formation. Front Neurol Neurosci. 2014;34:6-17. doi: 10.1159/000360925. Epub 2014 Apr 16. PMID 24777126
- [Result] Anderson JE, Trujillo M, McElroy T, Groves T, Alexander T, Kiffer F, Allen AR. Early Effects of Cyclophosphamide, Methotrexate, and 5-Fluorouracil on Neuronal Morphology and Hippocampal-Dependent Behavior in a Murine Model. Toxicol Sci. 2020 Jan 1;173(1):156-170. doi: 10.1093/toxsci/kfz213. PMID 31651976
- [Result] Yap NY, Toh YL, Tan CJ, Acharya MM, Chan A. Relationship between cytokines and brain-derived neurotrophic factor (BDNF) in trajectories of cancer-related cognitive impairment. Cytokine. 2021 Aug;144:155556. doi: 10.1016/j.cyto.2021.155556. Epub 2021 May 10. PMID 33985854
- [Result] Sommer C, Kress M. Recent findings on how proinflammatory cytokines cause pain: peripheral mechanisms in inflammatory and neuropathic hyperalgesia. Neurosci Lett. 2004 May 6;361(1-3):184-7. doi: 10.1016/j.neulet.2003.12.007. PMID 15135924
- [Result] Werida RH, Elshafiey RA, Ghoneim A, Elzawawy S, Mostafa TM. Role of alpha-lipoic acid in counteracting paclitaxel- and doxorubicin-induced toxicities: a randomized controlled trial in breast cancer patients. Support Care Cancer. 2022 Sep;30(9):7281-7292. doi: 10.1007/s00520-022-07124-0. Epub 2022 May 21. PMID 35596774
- [Result] Odabasoglu F, Halici Z, Aygun H, Halici M, Atalay F, Cakir A, Cadirci E, Bayir Y, Suleyman H. alpha-Lipoic acid has anti-inflammatory and anti-oxidative properties: an experimental study in rats with carrageenan-induced acute and cotton pellet-induced chronic inflammations. Br J Nutr. 2011 Jan;105(1):31-43. doi: 10.1017/S0007114510003107. Epub 2010 Nov 15. PMID 21073761
- [Result] Biewenga GP, Haenen GR, Bast A. The pharmacology of the antioxidant lipoic acid. Gen Pharmacol. 1997 Sep;29(3):315-31. doi: 10.1016/s0306-3623(96)00474-0. PMID 9378235
- [Result] Haghighatdoost F, Hariri M. The effect of alpha-lipoic acid on inflammatory mediators: a systematic review and meta-analysis on randomized clinical trials. Eur J Pharmacol. 2019 Apr 15;849:115-123. doi: 10.1016/j.ejphar.2019.01.065. Epub 2019 Feb 2. PMID 30721699
- [Result] Al-Majed AA, Gdo AM, Al-Shabanah OA, Mansour MA. Alpha-lipoic acid ameliorates myocardial toxicity induced by doxorubicin. Pharmacol Res. 2002 Dec;46(6):499-503. doi: 10.1016/s1043661802002311. PMID 12457622
- [Result] Aliomrani M, Mesripour A, Mehrjardi AS. Creatine and Alpha-Lipoic Acid Antidepressant-Like Effect Following Cyclosporine A Administration. Turk J Pharm Sci. 2022 Apr 29;19(2):196-201. doi: 10.4274/tjps.galenos.2021.27217. PMID 35510329
- [Result] Costa DSJ, Loh V, Birney DP, Dhillon HM, Fardell JE, Gessler D, Vardy JL. The Structure of the FACT-Cog v3 in Cancer Patients, Students, and Older Adults. J Pain Symptom Manage. 2018 Apr;55(4):1173-1178. doi: 10.1016/j.jpainsymman.2017.12.486. Epub 2017 Dec 30. PMID 29291932
- [Result] Limpawattana P, Manjavong M. The Mini-Cog, Clock Drawing Test, and Three-Item Recall Test: Rapid Cognitive Screening Tools with Comparable Performance in Detecting Mild NCD in Older Patients. Geriatrics (Basel). 2021 Sep 16;6(3):91. doi: 10.3390/geriatrics6030091. PMID 34562992
- See also: a full description of the MMSE — http://www.healthdirect.gov.au/mini-mental-state-examination-mmse